CLINICAL TRIAL: NCT06596226
Title: Evaluating The Efficacy of Pathways Parent-Mediated Intervention's Mutual Gaze Protocol on Social Skills in Young Children Suspected of Having Autism: A Randomized Control Trial
Brief Title: Evaluating Pathways Mutual Gaze Protocol on Social Skills in Young Children Suspected of Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Texas Higher Education Coordinating Board (Other Government)
Responsible Party: Principal Investigator, Pamela Rollins, Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTD IRB 24-804
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Autism
Keywords: Autism Intervention; Social development; Social communication
MeSH Terms: conditions — Autistic Disorder; Communication

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pathways with a Mutal Gaze Protocol (Experimental): 12 90-minute sessions (or 15 weeks, whichever comes first) of Pathways manualized Naturalistic Developmental Behavioral Intervention (NDBI) parent-mediated intervention (research version). Pathways uses a coaching model.
  Interventions: Behavioral: Pathways Parent Mediated Intervention
- Pathways without Mutual Gaze Protocol (Active Comparator): 12 90-minute sessions (or 15 weeks, whichever comes first) of Pathways manualized Naturalistic Developmental Behavioral Intervention (NDBI) parent-mediated intervention (research version) without the Mutual Gaze protocol. Pathways uses a coaching model.
  Interventions: Behavioral: Pathways Parent Mediated Intervention without Mutual Gaze

INTERVENTIONS:
Behavioral: Pathways Parent Mediated Intervention — Pathways-trained research clinicians will conduct 90-minute weekly coaching sessions with caregivers in the family's home or other convenient location. Caregivers will receive a written version of the program manual. Sessions will review information about social communication, infusing mutual gaze in social sensory routines, and using naturalistic developmental behavioral strategies. Interventionists will demonstrate intervention strategies and provide caregivers with practice feedback and self-reflection.
  Arms: Pathways with a Mutal Gaze Protocol
Behavioral: Pathways Parent Mediated Intervention without Mutual Gaze — Pathways-trained research clinicians will conduct 90-minute weekly coaching sessions with caregivers in the family's home or other convenient location. Caregivers will receive a written version of the program manual. Sessions will review information about social communication, social sensory routines, and naturalistic developmental behavioral strategies described in the program manual. Interventionists will demonstrate intervention strategies and provide caregivers with practice feedback and self-reflection.
  Arms: Pathways without Mutual Gaze Protocol

SUMMARY:
Purpose of the Study: The goal of this clinical trial is to find out if a technique called the "mutual gaze procedure," used in Pathways Early Intervention (Pathways), is the key to helping improve social communication, language, and everyday skills in young children (16-30 months old) who are at high risk for autism, particularly those from diverse cultural and language backgrounds.

What Will Happen: Researchers will compare two versions of the Pathways Intervention:

* Version 1: Includes mutual gaze strategies.
* Version 2: Does not include mutual gaze strategies.

What to Expect: Participants will:

* Attend 12 sessions of Pathways Intervention, each lasting 1.5 hours (or 15 weeks if there are cancellations).
* Come to the clinic for a developmental check-up three times: before starting Pathways, right after completing Pathways, and three months after finishing Pathways.

DETAILED DESCRIPTION:
Purpose of the Study: The primary goal of this clinical trial is to evaluate whether a parent-mediated treatment can improve social communication, language, and adaptive functioning in 16-30-month-old children from diverse cultural and language backgrounds who are at high risk for autism (referred to as children with social challenges).

Study Design:

* Study Phase: N/A
* Intervention Model: Participants are assigned to one of two groups in parallel.

Study Description:

* Participants: 80 children aged 16-30 months who show social communication challenges and are at high risk for autism will be randomly assigned to one of two groups:

  1. Group 1: Pathways Intervention with mutual gaze strategies.
  2. Group 2: Pathways Intervention without mutual gaze strategies.
* Intervention Sessions: Participants will attend 12 sessions, each lasting 1.5 hours, over approximately 15 weeks (allowing for possible cancellations) of parent-mediated intervention in their homes or another convenient location.

Assessments: To track progress and evaluate long-term effects, participants will undergo several culturally and linguistically appropriate assessments at three time points:

1. Baseline: Within two weeks before starting the intervention.
2. Post-Intervention: Within two weeks after completing the intervention.
3. Three-Month Follow-Up: 12-15 weeks after completing the intervention.

Each evaluation will take around two hours and will include:

* Child Assessments:

  * Mullen Scale of Early Learning (MSEL): Assesses general developmental age (administered only at baseline).
  * Communication and Symbolic Behavior Scales-Developmental Profile (CSBS-DP): Evaluates social communication.
  * EarliPointTM: Measures social, verbal, and nonverbal cognition.
* Caregiver Questionnaires:

  * Vineland Adaptive Behavior Scales, Third Edition (VABS-III): Assesses adaptive functioning.
  * PhenX Toolkit Core Measures: Collects family and child demographic information, including parents' and grandparents' place of birth (administered only at baseline).

The CSBS-DP and VABS-III have been validated as appropriate measures for determining meaningful changes in children with or at high risk for autism, based on previous research

ELIGIBILITY:
Inclusion Criteria:

* Children must be between 16-30 months old at the start of the study;
* Children must receive social disability index of 7 or lower on the EarliPointTM assessment with a researcher (i.e., human) confirming social challenges are present;
* Parents must report no other known neurological or genetic concerns or disorders
* Parents must be fluent in English
* Parents must live within a 30-mile radius of the Callier Center Dallas.

Exclusion Criteria:

* Children younger than 16 months or older than 30 months at the start of the study
* Children who are not at high risk for autism based on an EarliPointTM assessment (with researcher confirmation of social challenges)
* Children whose parents report they have any other known neurological or genetic concerns or disorders;
* Children whose parents are not fluent in English.

Ages: 16 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Improved Social skills | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Assessors blind to group assignment will evaluate each child for social skills using the EarliPointTM The EarliPointTM is an FDA-authorized eye-tracking tool that uses artificial intelligence (AI) eye-tracking technology to assess social disability in children between 16 and 30 months by measuring the number of social interactions a child observes on the portable eye-tracking screen. EarliTech will be used to measure improved social skills. There are 2 different EarliTech Scores: social disability and Verbal and nonverbal. Social disability scores range from -15 to +25, higher scores indicate better ability. Verbal and nonverbal scores range from 0-90, high scores indicate better ability.
Improved Social Communication Skills | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  Change in the raw scores obtained on the social, speech and symbolic composite of The Communication and Symbolic Behavior Scales- Developmental Profile (CSBS-DP) will be measured. Raw scores for the social, speech and symbolic composite range from 0-64, 0-54 and 0-53 respectively, 0 being the worst score. The CSBS-DP is a direct assessment of early social communication.
Change in Adaptive Functioning | At baseline (i.e., within two weeks prior to the start of intervention); Post-intervention (i.e., within two weeks after completing the intervention); At three-month follow-up
  The Vineland II is a standardized parent interview to assess adaptive functioning. Change in raw scores obtained on Vineland Adaptive Behavior Scales, Second Edition (Vineland II) will be measured. The Vineland II has 4 domains - Communication, Daily Living, Social Skills and Relationships, Physical Activity. The raw scores for these domains range from 0-252, 0-286, 0-224, 0-154 respectively (lower scores being worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Rollins, EdD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Considering reporting the collected data to the National Institute of Mental Health Data Archive (NDA). NDA provides a robust system for defining data dictionaries and metadata for all datasets, and the uploaded data itself will be in delimited plain text format. The shared data will include demographic data and measures administered to participants, as well as analyzed data.

REFERENCES:
- [Background] Anagnostou E, Jones N, Huerta M, Halladay AK, Wang P, Scahill L, Horrigan JP, Kasari C, Lord C, Choi D, Sullivan K, Dawson G. Measuring social communication behaviors as a treatment endpoint in individuals with autism spectrum disorder. Autism. 2015 Jul;19(5):622-36. doi: 10.1177/1362361314542955. Epub 2014 Aug 5. PMID 25096930
- [Background] (Anagnostou et al., 2015; Chatham et al., 2018; McCracken et al., 2021).
- [Background] Chatham CH, Taylor KI, Charman T, Liogier D'ardhuy X, Eule E, Fedele A, Hardan AY, Loth E, Murtagh L, Del Valle Rubido M, San Jose Caceres A, Sevigny J, Sikich L, Snyder L, Tillmann JE, Ventola PE, Walton-Bowen KL, Wang PP, Willgoss T, Bolognani F. Adaptive behavior in autism: Minimal clinically important differences on the Vineland-II. Autism Res. 2018 Feb;11(2):270-283. doi: 10.1002/aur.1874. Epub 2017 Sep 21. PMID 28941213
- [Background] McCracken JT, Anagnostou E, Arango C, Dawson G, Farchione T, Mantua V, McPartland J, Murphy D, Pandina G, Veenstra-VanderWeele J; ISCTM/ECNP ASD Working Group. Drug development for Autism Spectrum Disorder (ASD): Progress, challenges, and future directions. Eur Neuropsychopharmacol. 2021 Jul;48:3-31. doi: 10.1016/j.euroneuro.2021.05.010. Epub 2021 Jun 19. PMID 34158222
- [Background] Mullen, E. M. (1995). Mullen Scales of Early Learning. American Guidance Service, Guilford Press.
- [Background] Wetherby, A., & Prizant, B. (2002). Communication and Symbolic Behavior Scales- Developmental Profile (1st normed ed.). Paul H. Brookes.
- [Background] Sparrow, S. S., Cicchetti, D. V., & Saulnier, C. A. (2016). Vineland Adaptive Behavior Scales, Third Edition (Vineland-3). Pearson.